CLINICAL TRIAL: NCT04446260
Title: A Phase 1 Multi-Country, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-A1811 in HER2 Expressing or Mutated Advanced Malignant Solid Tumor Subjects
Brief Title: A Study of SHR-A1811 in Subjects With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-I-101
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose escalation (Experimental)
  Interventions: Drug: SHR-A1811
- Part 2 PK expansion (Experimental)
  Interventions: Drug: SHR-A1811
- Part 3 Indication expansion (Experimental)
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — be administered via intravenous (IV) infusion

SUMMARY:
This is an open-label, two-part study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of SHR-A1811 and preliminary anti-tumor efficacy in HER2 expressing or mutated advanced malignant solid tumor subjects.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/unresectable or metastatic solid tumor with HER2 expression or mutation that is refractory to or intolerable with standard treatment, or for which no standard treatment is available
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* LVEF ≥ 50% by either ECHO or MUGA
* Has adequate renal and hepatic function
* Female subjects agree not to be pregnant or lactating from beginning of the study screening until 6 months after receiving the last treatment

Exclusion Criteria:

* History of clinically significant lung diseases (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or suspected to have these diseases by imaging at screening period
* Known hereditary or acquired bleeding and thrombotic tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From Day1 to 90 days after last dose
  Frequency and seriousness of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
PK parameter: Tmax of SHR-A1811 | Through study completion, an average of 1 year
  Time to maximal concentration (Tmax) of SHR-A1811
PK parameter: Cmax of SHR-A1811 | Through study completion, an average of 1 year
  Maximal concentration (Cmax) of SHR-A1811
PK parameter: AUC0-t of SHR-A1811 | Through study completion, an average of 1 year
  AUC computed from time zero to the time of the last quantifiable concentration (AUC0-t) of SHR-A1811
Immunogenicity of SHR-A1811 | Through study completion, an average of 1 year
  Including anti-drug antibody and/or neutralizing antibody
Tumor response using RECIST 1.1 | From first dose to disease progression or death, whichever comes first, up to 30 months
  RECIST=Response Evaluation Criteria in Solid Tumors Assessment of tumor response until disease progression or death to evaluate the efficacy of SHR-A1811 up to 30 months

CONTACTS AND LOCATIONS:
Locations (35):
- United States (3):
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Greenville Hospital System, Greenville, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
- Australia (5):
  - Macquarie University Hospital, Macquarie, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Alfred Hospital, Melbourne
- China (21):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fujian, Fuzhou
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan cancer Hospital, Zhengzhou, Henan
  - Zhongnan hospital of Wuhan university, Wuhan, Hubei
  - Hubei cancer hospital, Wuhan, Hubei
  - Xiangya hospital central south university, Changsha, Hunan
  - Hunan cancer hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shengjing Hospital of China medical university, Shengyang, Liaoning
  - Fudan University Shanghai cancer center, Shanghai, Shanghai Municipality
  - Fudan Unversity Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiao Tong University School of Medicine Renji Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin medical university cancer institute&hoospital, Tianjin, Tianjin Municipality
  - The second affiliated hospital Zhejiang university school of medicine, Hangzhou, Zhejiang
  - Zhejiang provincial people's hospital, Hangzhou, Zhejiang
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao H, Yan M, Tong Z, Wu X, Ryu MH, Park JJ, Kim JH, Zhong Y, Zhao Y, Voskoboynik M, Yin Y, Liu K, Kaubisch A, Liu C, Zhang J, Wang S, Im SA, Ganju V, Barve M, Li H, Ye C, Roy AC, Bai LY, Yen CJ, Gu S, Lin YC, Wu L, Bao L, Zhao K, Shen Y, Rong S, Zhu X, Song E. Safety, Efficacy, and Pharmacokinetics of SHR-A1811, a Human Epidermal Growth Factor Receptor 2-Directed Antibody-Drug Conjugate, in Human Epidermal Growth Factor Receptor 2-Expressing or Mutated Advanced Solid Tumors: A Global Phase I Trial. J Clin Oncol. 2024 Oct 10;42(29):3453-3465. doi: 10.1200/JCO.23.02044. Epub 2024 Jun 20. PMID 38900984